CLINICAL TRIAL: NCT01143961
Title: Measurement of Changes in Ventilation and Catheter Placement During Non-directed Bronchoalveolar Lavage Using Electrical Impedance Tomography With and Without a One-way Valve
Brief Title: Bedside Measurement of Ventilation With or Without a One-way Valve During Lung Lavage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09/MRE09/54
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2010-02

CONDITIONS: Intensive Care
Keywords: Positive pressure ventilation; Electrical impedance tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBL with one-way valve (Experimental): NBL performed with one-way valve in ventilator circuit during procedure
  Interventions: Device: CSC100 - Verso airway access adapter CareFusion
- Standard NBL (No Intervention): Performance of standard NBL with recording of changes in regional ventilation by electrical impedance tomography

INTERVENTIONS:
Device: CSC100 - Verso airway access adapter CareFusion — Following randomisation patients will have a one-way valve inserted into the ventilator circuit (CSC100 - Verso airway access adapter CareFusion) prior to a non-directed bronchoalveolar lavage (NBL) being performed. Changes in regional ventilation will be recorded by electrical impedance tomography during the NBL. Recordings of ventilation will take place for upto four hours. One-way valve will stay in place until ventilator circuit is changed.
  Other Names: One-way adapter valve
  Arms: NBL with one-way valve

SUMMARY:
Surveillance of the lungs for bacteria is routinely undertaken in artificially ventilated patients as these individuals are at high risk of developing pneumonia. Knowledge of the types of bacteria present allows the rapid treatment with the correct antibiotics if a pneumonia develops. Surveillance is undertaken using a technique called non-directed bronchoalveolar lavage (NBL), which can be performed by the bedside nurse. This involves suctioning some of the lung secretions into a sample pot and sending it to the microbiology laboratory to identify any bacteria present. When this procedure is performed there is some collapse of the lung due to escaping gas. The purpose of this study is:

1. To use a non-invasive imaging technique known as electrical impedance tomography (EIT) to measure the amount of lung collapse during an NBL. Half of the patients in the study will have a one-way adapter valve connected to the breathing circuit. This adapter is designed to make the insertion of a suction catheter easier and prevent the loss of gas.
2. Look at which region of the lung the sample is being collected from as the suction tube used to take the samples may pass into either the left or right lung.

EIT is a simple non-invasive technique which has been in use for many years. It uses pairs of electrodes around the chest through which imperceptible currents are passed. A computer shows an image of which parts of the lungs have the most or least air in them. This has the advantage over other imaging techniques in critical care that it does not use radiation and gives a real time picture at the bedside of the variations in ventilation throughout the lungs.

DETAILED DESCRIPTION:
This study has two objectives. The first is to measure changes in lung ventilation using EIT during the performance of an NBL with and without a one-way adapter valve attached to the catheter mount. This will be done by randomising half of the patients to having the one-way adapter valve attached to the catheter mount. Assignment will be by randomisation.

The second objective of the study is to locate the placement of catheter tips during the performance of NBLs, using electrical impedance tomography.

Equipment: A sixteen-electrode single frequency electrical impedance tomography device with on-line image analysis (CareFusion). One-way adapter valves which attach to the catheter mount (CareFusion).

Study Population: Critically ill adult patients admitted to the intensive care unit at the University Hospital of Wales Cardiff in whom NBLs are performed as part of their routine care.

Recruitment: All patients satisfying inclusion and exclusion criteria, admitted to the adult ICU at the University Hospital of Wales from the start date of the study will be considered eligible for recruitment. Patients identified by the duty consultant will be notified to the research team. Patients will be randomly allocated to have NBLs performed with or without the one-way valve attached to the catheter mount.

Since this is an observational pilot study a minimum of fifty patients will be identified.

Interventions: The second cohort of patients will have NBLs performed with the one-way adapter connected to the catheter mount, otherwise there will be no change will be made to the normal standard of care.

Method: Following cleaning of the skin with alcohol wipes sixteen ECG electrodes will be placed equidistantly from one another midway between sternum and umbilicus. A reference electrode will be placed on the right hand side of the chest. NBLs will be undertaken according to routine standards of care. In brief, this involves pre-oxygenating the patient, and inserting a suction catheter attached to a 20ml saline filled syringe through the catheter mount (25 patients) or adapter with one-way valve connected to the catheter mount (25 patients) until resistance is met. The saline is instilled and then slowly withdrawn to obtain a sample. Since saline is conductive, instillation results in a change in local impedance which is detected by the array of electrodes. The image obtained will identify into which region of the lung the catheter is placed. Any changes in the gas content of lung (due to loss of PEEP) will be manifest as changes in lung impedance and reflects a change in regional ventilation. NBLs are undertaken when clinically indicated and patients may have more than one recoding undertaken up to a maximum of three times.

Collection of other data: Baseline demographics of patients will be recorded, including age, sex, APACHE II score, co-morbidities, diagnosis, days from hospital admission. Ventilator settings - mode, inspired oxygen fraction, tidal and minute ventilation, compliance, PEEP and mean airway pressure will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years
* Patients in whom an NBL is indicated as part of standard treatment
* Patient on mechanical ventilation with PEEP

Exclusion Criteria:

* NBL contraindicated
* Age <18 years
* Patient not on mechanical ventilation with PEEP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Measure changes in lung ventilation using EIT during the performance of an NBL with and without a one-way adapter valve attached to the catheter mount. | Up to 4 hours

SECONDARY OUTCOMES:
Locate the placement of catheter tips during the performance of NBLs, using electrical impedance tomography | Up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Matt P Wise, DPhil, Principal Investigator — University Hospital of Wales Cardiff & Vale University Health Board
Locations (1):
- Adult Critical Care, University Hospital of Wales, Cardiff, South Glamorgan, United Kingdom